CLINICAL TRIAL: NCT02395055
Title: Single Center Comparative Double Blind Randomized Clinical Study of Pharmacokinetics, Tolerance and Safety of Single Subcutaneous Injection of BCD-057 (JSC "BIOCAD", Russia) and Humira in Healthy Volunteers
Brief Title: Comparative Clinical Study of Pharmacokinetics, Tolerance and Safety of BCD-057 and Humira in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Biocad (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: BCD-057-1
Record Dates: First submitted 2015-03-16; First posted 2015-03-20 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2021-11-05 (Actual); Status verified 2021-10

CONDITIONS: Healthy
MeSH Terms: interventions — Adalimumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- BCD-057 group (Experimental): BCD-057 (adalimumab) at a dose of 40 mg, administered as a single subcutaneous injection, which will be performed on week 0.
  Interventions: Drug: Adalimumab (BCD-057)
- Humira group (Active Comparator): Humira (adalimumab) at a dose of 40 mg, administered as a single subcutaneous injection, which will be performed on week 0.
  Interventions: Drug: Adalimumab (Humira)

INTERVENTIONS:
Drug: Adalimumab (BCD-057) — Adalimumab is a monoclonal antibody against tumor necrosis factor alpha
  Other Names: BCD-057; Humira; Trudexa
  Arms: BCD-057 group
Drug: Adalimumab (Humira) — Adalimumab is a monoclonal antibody against tumor necrosis factor alpha
  Other Names: Trudexa
  Arms: Humira group

SUMMARY:
This clinical study is a phase 1 study which carried out to establish the pharmacokinetic equivalence and equal safety and tolerability profile of BCD-057 (adalimumab biosimilar candidate manufactured by CJSC BIOCAD, Russia) and Humira when used as a single subcutaneous injection in healthy volunteers.

DETAILED DESCRIPTION:
This is single center comparative double blind randomized clinical study of pharmacokinetics, tolerance and safety of single subcutaneous injection of BCD-057 (CJSC BIOCAD, Russia) and Humira in healthy volunteers. The purpose of the study is to demonstrate that BCD-057 is equivalent to Humira in terms of pharmacokinetics, tolerability and safety after single subcutaneous injection in healthy volunteers.

The study will enroll 94 healthy volunteers, who will be randomized into 2 groups (1:1 ratio): volunteers from the first group will receive BCD-057; volunteers from the second group will receive Humira. Both study and reference drug will be used at the standard dose of 40 mg.

ELIGIBILITY:
Inclusion Criteria:

* subject has provided informed consent;
* male gender;
* 18 - 45 years of age inclusively;
* a body mass index (BMI) between 18,5 and 30 kg/m2;
* absence of clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality at screening or/and in anamnesis;
* parameters of complete blood count, blood biochemistry and urinalysis do not exceed reference values, which are used at Study site laboratory. Evaluation of required laboratory parameters must be performed within 14 days before randomization;
* normal hemodynamic parameters: systolic BP 100 - 139 mm Hg, diastolic BP - 60 - 90 mm Hg, heart rate - 60 - 90 b/min;
* ECG results are normal for this age group;
* absence of chronic infections (HIV, syphilis, hepatitis В or С) and chronic inflammation;
* absence of active or latent tuberculosis;
* absence of infections within 4 weeks before randomization;
* absence of mental disorders or other conditions, which may affect the ability of participant to follow Protocol;
* health well-being (by volunteer's opinion) for at least 30 days before randomization;
* ability to follow Protocol procedures;
* consent of volunteers and their sexual partners with childbearing potential to use adequate contraception during screening period and the main study part;
* absence of alcohol or drug addiction signs (incl. history of such addiction);
* consent not to consume alcohol within 24 hours before SC injection of BCD-057/Humira and not to use more than 10 units of alcohol per week during the study (1 alcohol unit is equal ½ l of beer (1 pint), or 200 ml of wine, or 50 ml alcohol)

Exclusion Criteria:

* history of adalimumab use or any other TNF inhibitors;
* known severe allergy (anaphylaxis or multidrug intolerance);
* known intolerance of monoclonal antibodies or any other excipients of BCD-057/Humira;
* major surgery within 30 days before ICF signing;
* presence of clinically significant hepatic, renal, gastrointestinal, cardiovascular, endocrine, respiratory, immunologic, hematologic, dermatologic, or neurologic abnormality at screening or/and in anamnesis.
* infections which required hospitalization, parenteral anti-infectives within 6 months before randomization;
* positive results of tests for HIV-1 and HIV-2 antibodies, positive Hbs-Ag, HBc IgM, total antibodies against HCV, positive results of RPR-test;
* more than 4 episodes of acute respiratory infection within 6 months before randomization;
* any malignancy (present or history);
* tuberculosis, including latent forms;
* shingles (present or history).
* history of seizures;
* any disorders or other conditions, which may affect pharmacokinetics of BCD-057/Humira (e.g. chronic liver diseases, chronic kidney diseases, cardiovascular disorders, lung disorders, endocrine diseases, etc.).
* use of systemic antimicrobial or antifungal medicines within 2 months before randomization;
* regular oral or parenteral use of any medicines, vitamins, biologically active additives within two weeks before signing of ICF;
* any use of medicines, vitamins, biologically active additives within 30 days before signing of ICF;
* use of medicines, which may influence on immunity within 30 days before signing of ICF;
* vaccination within 4 weeks prior randomization;
* smoking of more than 10 cigarettes per day;
* use of alcohol, which exceeds 10 units per week (1 alcohol unit is equal ½ l of beer (1 pint), or 200 ml of vine, or 50 ml alcohol). History of alcohol or drug addiction;
* donation of more than 450 ml of blood or plasma within 2 months prior randomization;
* simultaneous participation in any other clinical trial, as well as former participation in other clinical trials within 3 months before this study initiation;
* previous participation in this study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 94 (Actual)
Dates: Start 2015-06; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Roman Ivanov, Phd, Study Chair — CJCS BIOCAD
Locations (1):
- LLC BioEk, Saint Petersburg, Russia

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | BCD-057 Group | Humira Group
Started | 47 | 47
Completed | 40 | 44
Not Completed | 7 | 3
Not completed — Withdrawal by Subject | 7 | 3

BASELINE CHARACTERISTICS:
Population: Population for all type of analysis included 84 patients who received at least one study drug injection.
Groups:
- Total: Total of all reporting groups
Arm/Group | BCD-057 Group | Humira Group | Total
Number analyzed (Participants) | 40 | 44 | 84
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 40 | 44 | 84
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 24.5 [22 to 30.5] | 25.5 [22 to 29] | 25 [22 to 30]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 40 | 44 | 84

OUTCOME MEASURES:

1. Primary Outcome: Maximum Concentration of Adalimumab After Single SC Injection of BCD-057/Humira
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Population: All patients who received one injection of adalimumab.
Measure: Median (Inter-Quartile Range); unit: ng/ml
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
ng/ml | 4426 [3524 to 5902] | 4522 [3546 to 5104]

2. Primary Outcome: Area Under the Plasma Concentration-time Curve From Zero (0) to Time Infinity
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Population: All patients who received adalimumab injection.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
(ng/ml)*hour | 2488188 [1809194 to 2827564] | 2272029 [1815831 to 2904679]

3. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Zero (0) Hours to 1680 Hours of Adalimumab After Single SC Injection of BCD-057/Humira.
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Population: All volunteers who received one adalimumab injection.
Measure: Median (Inter-Quartile Range); unit: (ng/ml)*hour
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
(ng/ml)*hour | 2488187 [1809193 to 2778993] | 2272029 [1815831 to 2858812]

4. Secondary Outcome: Time to Reach Maximum Concentration of Adalimumab After Single Subcutaneous Injection of BCD-057/Humira
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
hours | 120 [96 to 192] | 108 [90 to 150]

5. Secondary Outcome: Half-life Period of Adalimumab After Single Subcutaneous Injection of BCD-057/Humira
Time Frame: 0, 6, 24, 48, 72, 96,120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
hours | 263.35 [194.65 to 351.61] | 269.68 [196.29 to 317.01]

6. Secondary Outcome: Volume of Distribution of Adalimumab After Single Administration of BCD-057/Humira
Time Frame: 0, 6, 24, 48, 72, 96,120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Measure: Median (Inter-Quartile Range); unit: ml/kg
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
ml/kg | 7165.85 [5105.07 to 8482.38] | 6622.06 [5637.07 to 7854.49]

7. Secondary Outcome: Clearance of Adalimumab After Single Subcutaneous Injection of BCD-057/ Humira
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Measure: Median (Inter-Quartile Range); unit: ml/(h*kg)
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
ml/(h*kg) | 16.08 [14.39 to 22.11] | 17.61 [13.99 to 22.04]

8. Secondary Outcome: Elimination Rate Constant of Adalimumab After Single Subcutaneous Injection of BCD-057/Humira
Time Frame: 0, 6, 24, 48, 72, 96, 120, 144, 168, 192, 336, 672, 1008, 1440, 1680 hours post-dose
Measure: Median (Inter-Quartile Range); unit: fraction of drug eliminated per hour
Arm/Group | BCD-057 Group | Humira Group
Number analyzed (Participants) | 40 | 44
fraction of drug eliminated per hour | 0.003 [0.002 to 0.004] | 0.003 [0.002 to 0.004]

ADVERSE EVENTS:
Time Frame: 70 days
Arm/Group | BCD-057 Group | Humira Group
Serious Adverse Events (participants affected / at risk) | 0/40 | 0/44
Other Adverse Events (participants affected / at risk) | 9/40 | 14/44
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | BCD-057 Group (N=40) | Humira Group (N=44)
Leucopenia (Blood and lymphatic system disorders) | 1 | 2
Neutropenia (Blood and lymphatic system disorders) | 2 | 1
Monocytosis (Blood and lymphatic system disorders) | 2 | 0
Monocytopenia (Blood and lymphatic system disorders) | 2 | 1
Hyperbilirubinemia (Hepatobiliary disorders) | 2 | 2
Elevated ALT (Hepatobiliary disorders) | 3 | 11
Elevated AST (Hepatobiliary disorders) | 3 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No